CLINICAL TRIAL: NCT02257762
Title: Efficacy of a Locally-Produced Multiple Micronutrient-Fortified Lipid-Based Nutrient Supplement (LNS) for Children Under Two Years in Cambodia
Brief Title: Efficacy of a Multiple Micronutrient-Fortified Lipid-Based Nutrient Supplement for Children Under Two in Cambodia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Institut de Recherche pour le Developpement, Cambodia (Other Government)
Collaborators: UNICEF (Other); Department of Fisheries Post-harvest Technologies and Quality Control (Other)
Responsible Party: Principal Investigator, Bindi Borg, PhD Candidate, University of Sydney
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: LNS-CAMB-INFANTS-EFF
Record Dates: First submitted 2014-10-02; First posted 2014-10-06 (Estimated); Last update posted 2016-09-15 (Estimated); Status verified 2016-09

CONDITIONS: Child Malnutrition
Keywords: Ready-to-use supplementary food (RUSF); Lipid-based nutrient supplement (LNS); Multiple micronutrients (MMN); Complementary feeding; Home fortification; Efficacy/impact; Infant and young child feeding (IYCF); Cambodia; Cluster randomised controlled trial
MeSH Terms: conditions — Child Nutrition Disorders; Tooth, Impacted

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Lipid-based nutrient supplement (LNS) (Experimental): LNS added to borbor, eaten over 6 months, age 6-12 months to age 11-17 months
  Interventions: Dietary Supplement: LNS
- Corn-soy blend ++ (CSB++) (Active Comparator): CSB++ porridge, eaten over 6 months, age 6-12 months to age 11-17 months
  Interventions: Dietary Supplement: Corn-soy blend ++ (CSB++)
- Sprinkles (Active Comparator): Sprinkles added to borbor, eaten over 6 months, age 6-12 months to age 11-17 months
  Interventions: Dietary Supplement: Sprinkles
- Control (No Intervention): Plain borbor and thereafter family foods, eaten over 6 months, age 6-12 months to age 11-17 months

INTERVENTIONS:
Dietary Supplement: LNS — Compact, paste-filled wafer snack containing fish, rice, soy, mungbeans, oil, sugar and multiple micronutrients
  Arms: Lipid-based nutrient supplement (LNS)
Dietary Supplement: Corn-soy blend ++ (CSB++) — Blended flour containing soy, corn, milk powder, oil, sugar and multiple micronutrients.
  Other Names: Supercereal Plus
  Arms: Corn-soy blend ++ (CSB++)
Dietary Supplement: Sprinkles — Multiple micronutrient powder packaged in sachet.
  Arms: Sprinkles

SUMMARY:
The purpose of this trial is to evaluate the efficacy of the LNS on children aged 6-17 months in preventing growth faltering and improving micronutrient status. The impact of product will be compared to Corn Soy Blend ++ (CSB++), Sprinkles, and to a control group consuming an unsupplemented diet, which is usually borbor at an early age, and thereafter, family foods.

DETAILED DESCRIPTION:
BACKGROUND:

In Cambodia, progress in combatting malnutrition has stalled. In 2010, 40% of all children under five (and 49% of 4-5 year-olds) were stunted, 11% were wasted, and 28% were underweight, indicating, respectively, chronic and acute malnutrition, and a combination of the two. Stunting is partially attributed to poor complementary feeding, which remains inadequate for achieving growth outcomes and micronutrient status.

Malnutrition can be prevented with supplementary foods. These foods usually contain a source of protein and lipids such as powered milk, soy or peanuts, and multiple micronutrients. They can be prepared as a fortified blended product, such as Corn-Soy Blend++ (CSB++), that is mixed with water to make a porridge, or ready-to-use supplementary foods (RUSFs). The latter are usually lipid-based nutrient supplements (LNSs) which are often pastes such as the peanut-based Plumpy'Nut™. These energy-dense supplementary foods contain both macro and micronutrients and are used to prevent and treat moderate acute malnutrition by promoting improved linear growth, weight gain and micronutrient status among children. Until recently, treatment of moderate acute malnutrition has relied on fortified blended products. The new RUSFs are also proving effective, as they are higher energy and have a longer shelf life, and since they require no preparation, are convenient. Another common nutrition intervention is multiple micronutrient supplements such as Sprinkles. These are individually-packed powders that can be added to food. However, micronutrients are more likely to achieve growth outcomes when they are combined with energy, for example, in lipid-based nutrient supplements and there is no evidence that micronutrient powders alone contribute to growth.

Until June 2014, the United Nations World Food Program (WFP) used CSB++ (now called Supercereal Plus) to treat and prevent moderate acute malnutrition in Cambodia. Sprinkles are also being distributed, though not widely, to prevent micronutrient deficiencies. These products that have been recently or are currently used are relatively expensive to procure and ship to Cambodia and in the case of Sprinkles, are not as effective as foods that contain macronutrients. Moreover, CSB++ was not very well accepted in practice, and WFP has phased it out. Therefore, UNICEF and the Cambodian Ministry of Health are looking for a locally-produced product containing macro and micronutrients to prevent growth faltering and improve micronutrient status in Cambodian children.

TRIAL DESIGN AND METHODOLOGY:

Therefore, this trial will evaluate the efficacy of the LNS on children aged 6-17 months in preventing growth faltering and improving micronutrient statu. The impact of product will be compared to CSB++, Sprinkles, and to a control group.

The trial is a prospective, cluster randomised, non-blinded controlled trial among infants 6-17 months of age. The trial aims to establish the superiority of the novel LNS, using CSB++ and Sprinkles as active comparators and the unimproved diet as a control. The allocation ratio is 1:1. The study will take place over 8 months.

The study will be conducted in 28 sites in peri-urban Phnom Penh. Infants aged 6-12 months will be recruited. Upon consent and enrolment, baseline data will be collected from the participants. This will include demographics, morbidity, anthropometry (weight, height, mid-upper arm circumference, skinfolds), haematological and stool samples, dietary data (breastfeeding, food frequency and dietary diversity). Data will be collected monthly, and haematological samples will be collected again at endline.

Participants will then be provided with a one month supply of the food to which their site has been allocated. Staff will explain how to prepare the food, how often it should be consumed, and who should consume it (i.e. subjects). Participants will be provided with food on a monthly basis. They will continue to consume the food over a six-month period, at which time endline data, including haematological samples, will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 6-12 months
* Normally nourished or only moderately malnourished (MUAC>115mm, WHZ score>-3)
* Have not received therapy for acute malnutrition within one month prior to presentation
* Healthy (no ill-health in past two weeks)
* Anaemia status - normal, mild or moderate
* No known food intolerances
* Informed signed consent of caregiver
* Caregivers are healthy

Exclusion Criteria:

* Children <6 months or >12mths
* Severely malnourished (MUAC< 115mm, WHZ score<3, bipedal pitting oedema).
* Have received therapy for acute malnutrition within one month prior to presentation
* Any medical complications at the recruitment time or illness requiring referral or clinic visit in past 2 weeks
* Severe anaemia (Hb<70g/l)
* Known intolerances
* No informed signed consent of caregiver

Ages: 6 Months to 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 487 (Actual)
Dates: Start 2016-02; Primary Completion 2016-10 (Estimated); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
Nutritional status | 6 months
  Weight-for-height (WHZ), length/height-for-age (L/HAZ), and weight-for-age (WAZ) calculated through monthly weight and height measurements

SECONDARY OUTCOMES:
Body composition | 6 months
  Triceps, biceps and/or subscapular skinfolds
Iron status | 6 months
  Analysis of haemoglobin (g/l), ferritin (µg/l), tranferrin receptor (mg/l), C reactive protein (mg/l), and alpha-1-acid glycoprotein (mg/l)

CONTACTS AND LOCATIONS:
Overall Officials: Frank T Wieringa, MD, PhD, Study Director — IRD; Bindi Borg, MA,PhD cand., Principal Investigator — University of Sydney
Locations (1):
- IRD Cambodia, Phnom Penh, Cambodia

REFERENCES:
- [Derived] Borg B, Sok D, Mihrshahi S, Griffin M, Chamnan C, Berger J, Laillou A, Roos N, Wieringa FT. Effectiveness of a locally produced ready-to-use supplementary food in preventing growth faltering for children under 2 years in Cambodia: a cluster randomised controlled trial. Matern Child Nutr. 2020 Jan;16(1):e12896. doi: 10.1111/mcn.12896. PMID 31885221
- [Derived] Borg B, Mihrshahi S, Griffin M, Sok D, Chhoun C, Laillou A, Berger J, Wieringa FT. Randomised controlled trial to test the effectiveness of a locally-produced ready-to-use supplementary food (RUSF) in preventing growth faltering and improving micronutrient status for children under two years in Cambodia: a study protocol. Nutr J. 2018 Mar 16;17(1):39. doi: 10.1186/s12937-018-0346-x. PMID 29548287